CLINICAL TRIAL: NCT00955318
Title: Phase 3 Study of KW-6500 (Safety Study for Long-Term Self-Administration at Home in Patients With Parkinson's Disease
Brief Title: Long-Term Safety Study of KW-6500 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6500-003
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- KW-6500 (Experimental)
  Interventions: Drug: KW-6500

INTERVENTIONS:
Drug: KW-6500 — Subcutaneous injection of 1to 6 mg of KW-6500 for the OFF state
  Other Names: Apomorphine hydroshloride (USAN)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of KW-6500 when administered as long-term subcutaneous self-injections in Parkinson's disease patients with motor response complications on levodopa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Patients who have Parkinson's disease
* Patients who have been on a stable regimen of levodopa plus at least one other antiparkinsonian agent and who have OFF state
* Patients who meet stage 4 or 5 while in the OFF state and stage 0 to 3 while in the ON state on the Modified Hoehn and Yahr Scale
* Patients who have experienced a 30% or more improvement in UPDRS partⅢ score when tested for responsiveness to levodopa during the baseline period
* Patients who have at least one OFF state per day
* Patients who can understand the expression of OFF state, ON state, and dyskinesia
* Patients or their families have a desire for self-injection of KW-6500

Exclusion Criteria:

* Patients with an illness of the cardiac, hematologic, hepatic, renal, pancreatic, metabolic, respiratory, gastrointestinal, endocrinologic, or neurologic system (excluding Parkinson's disease)
* Patients with orthostatic hypotension
* Patients with a history of intolerance to morphine or its derivatives, sulfur, sulfur-containing pharmaceutical products, or sulfite
* Patients with a history of malignant syndrome
* Patients with a diagnosis of cancer or evidence of continued disease
* Patients who do not test negative in the direct Coombs' test
* Pregnant or lactating women, women who are planning to have children, women who test positive in the pregnancy test, or women who cannot adhere to a reliable method of contraception
* Patients who have received MAO inhibitors except selegiline
* Patients with a history of mental disease (excluding psychiatric symptoms associated with Parkinson's disease)
* Patients with a Mini-Mental State Examination (MMSE) score of 23 or less
* Patients who are taking antipsychotics or central dopamine antagonists (excluding domperidone)
* Patients who are receiving methyldopa or 5-HT3 receptor antagonists
* Patients who are receiving reserpine or papaverine
* Patients who have had a neurosurgical operation for Parkinson's disease
* Patients who have had transcranial magnetic stimulation
* Patients with a history of drug or alcohol abuse or dependence

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events after administration of KW-6500 | From first administration of study drug through Study Week 52
Time to expression of the ON state, continuous time of the ON state, raw score change and percent score change in Unified Parkinson's Disease Rating Scale (UPDRS) part III, response ratio, and UPDRS part II score | From first administration of study drug through Study Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan